CLINICAL TRIAL: NCT01443325
Title: Lidocaine Patch for Treatment of Persistent Inguinal Postherniorrhaphy Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Joakim Bischoff, Research fellow, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2-2011-051
Record Dates: First submitted 2011-09-26; First posted 2011-09-29 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Inguinal Pain
Keywords: Persistent Postherniorrhaphy inguinal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lidocaine patch (Experimental)
  Interventions: Drug: lidocaine patch

INTERVENTIONS:
Drug: lidocaine patch — 1 patch for 12 hours within each 24 hours period
  Other Names: versatis

SUMMARY:
In the present placebo-controlled cross-over study the researchers intend to investigate analgesic and sensory effects of a lidocaine patch in patients with severe persistent inguinal post-herniorrhaphy pain.

ELIGIBILITY:
Inclusion Criteria:

* Males > 18 yrs
* ASA (American Society´s of Anesthesiology´s classification) scores I-III, with severe Pain for more than six months and with average daily pain intensities (numerical rating scale [NRS] 0-10 points) during rest or during movement > 6.

Exclusion Criteria:

* History of an allergic reaction or intolerance to amide local anesthetics or vehicle ingredients in the patches
* Use of class I antiarrhythmic drugs (e.g., tocainide and mexiletine)
* Severe cardiac impairment, e.g., NYHA (New York Heart Association) Class ≥ III
* Inflamed or injured skin at the application site
* Known severe hepatic disorder (Child-Pugh score > 6)
* Known severe renal impairment, (creatinine clearance < 30 mL/min)
* Signs of cognitive impairment or known drug or ethanol abuse during the last 2 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
pain reduction with lidocaine patch | assessed the last three days in each treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark